CLINICAL TRIAL: NCT03556501
Title: Comparative Registry of Structural Features of Pancreatic Collections Found on Cross Sectional Imaging
Brief Title: Imaging Modalities for Pancreatic Collections
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment numbers - participants are no longer being examined
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0228
Record Dates: First submitted 2018-04-24; First posted 2018-06-14 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Pancreas Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopy — Purpose of this study is to create a prospective registry of patients with pancreatic collections and their imaging studies

SUMMARY:
The purpose of this project is to provide appropriate administrative and technical supports for the warehousing and use of imaging data in pancreatic necrosis data for research purposes.

DETAILED DESCRIPTION:
The aim of this study is to create a prospective registry of patients with pancreatic collections and their imaging studies (including CT, MRI, EUS, and direct endoscopic visualization) to compare these techniques, develop standardized methods for analyzing these imaging studies, and use this information to enhance management of patients with pancreatic collections. There is very limited published literature on these peripancreatic lesions that compares all three of these modalities and thus we aim to study it in detail.

ELIGIBILITY:
Inclusion Criteria:

* patients who are known to have a pancreatic fluid collection after an episode of acute pancreatitis
* age greater than 18 years

Exclusion Criteria:

* pregnant woman
* age <18 years
* prisoners
* other institutionalized individuals
* patients who are decisionally impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at Northshore-LIJ being evaluate by the gastroenterology service
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
to define severity of pancreatitis as mild, moderate, severe; based on amount of debris in the pancreatic lesion (mild: < 30% debris, moderate: 30-50% debris, severe: >50% debris) | one year
  Pancreatic lesions will be evaluated using CT, MRI, EUS, endoscopy to assess for severeity based on amount of debris in the pancreatic lesion

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Trindade, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Hospital, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Bollen TL, Singh VK, Maurer R, Repas K, van Es HW, Banks PA, Mortele KJ. A comparative evaluation of radiologic and clinical scoring systems in the early prediction of severity in acute pancreatitis. Am J Gastroenterol. 2012 Apr;107(4):612-9. doi: 10.1038/ajg.2011.438. Epub 2011 Dec 20. PMID 22186977
- [Background] Singh VK, Bollen TL, Wu BU, Repas K, Maurer R, Yu S, Mortele KJ, Conwell DL, Banks PA. An assessment of the severity of interstitial pancreatitis. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1098-103. doi: 10.1016/j.cgh.2011.08.026. Epub 2011 Sep 3. PMID 21893128
- [Background] Tyberg A, Karia K, Gabr M, Desai A, Doshi R, Gaidhane M, Sharaiha RZ, Kahaleh M. Management of pancreatic fluid collections: A comprehensive review of the literature. World J Gastroenterol. 2016 Feb 21;22(7):2256-70. doi: 10.3748/wjg.v22.i7.2256. PMID 26900288